CLINICAL TRIAL: NCT00720681
Title: Plating of Acute Humeral Diaphyseal Fractures Via an Anterior Lateral Approach in Multiple Trauma Patients.
Brief Title: Plating of Humeral Shaft Fractures in Multiple Trauma Patients.
Acronym: HUMERUS
Status: Completed | Type: Observational
Sponsor: OhioHealth (Other)
Collaborators: Orthopaedic Trauma and Reconstructive Surgery (Unknown)
Responsible Party: Principal Investigator, Bruce French, Chief, OrthopedicTrauma, OhioHealth
Other Study IDs: 08-0014
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Humeral Fractures; Multiple Trauma
MeSH Terms: conditions — Humeral Fractures; Multiple Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to review our experience with the operative management of acute diaphyseal fractures of the humerus via an anterolateral approach with the use of small fragment fixation at a Level I, urban, trauma center. We will report our clinical and radiographic results, complication rate and final range of motion. A standardized outcome measurement (DASH) will be reported. Muscle recovery of the triceps and biceps will be evaluated by a standard protocol, accomplished with the assistance of a licensed physical therapist. We hypothesize that open reduction and internal fixation of humeral diaphyseal fractures via an antero-lateral approach with the use of small fragment fixation is a safe and efficacious way to treat multiple trauma patients with these injuries.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* patients with past (acute) traumatic humeral shaft fracture(s) treated with open reduction and internal fixation (ORIF)
* patients for whom the above fracture has healed
* patients willing and able to provide informed consent and able to participate in study procedures

Exclusion Criteria:

* patients with known pathological fractures
* patients with metabolic bone disease
* patients with humeral head or inter-articular surface fractures, or other upper extremity fractures
* patients with previous humeral surgery (i.e. rotator cuff, biceps tendon, etc.)
* patients with neurologic injury to upper extremities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated by our practice for diaphyseal fracture of the humerus after multiple trauma.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2008-08; Primary Completion 2009-06 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
DASH (Disabilities of the Arm, Shoulder and Hand) Score | At Enrollment
Strength of injured arm compared to uninjured arm | At enrollment
Range of motion in injured arm compared to uninjured arm | At enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Bruce French, M.D., Principal Investigator — Grant Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Idoine JD 3rd, French BG, Opalek JM, DeMott L. Plating of acute humeral diaphyseal fractures through an anterior approach in multiple trauma patients. J Orthop Trauma. 2012 Jan;26(1):9-18. doi: 10.1097/BOT.0b013e318214ebd5. PMID 21577147